CLINICAL TRIAL: NCT05658107
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Intravenous Doses of BI 765423 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Different Doses of BI 765423 Are Taken up in the Body of Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1493-0007; 2022-002501-18 (EudraCT Number)
Record Dates: First submitted 2022-12-13; First posted 2022-12-20 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 765423 treatment group (Experimental): BI 765423
  Interventions: Drug: BI 765423
- Placebo group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 765423 — BI 765423
  Arms: BI 765423 treatment group
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 765423 in healthy male subjects following intravenous administration of single rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male subjects who are willing to use condoms to prevent unintended exposure of their partner (both, male and female) from time point of administration of trial medication until completion of the trial. Male subjects with female partners must meet one of the following criteria for a highly effective contraception from at least screening until at least end-of-trial visit:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal) by female Women of child-bearing potential (WOCBP) partner, plus condom in male subject
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants) by female WOCBP partner, plus condom in male subject
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS) by female WOCBP partner, plus condom in male subject
  * Male subject is vasectomised (vasectomy at least 1 year prior to enrolment) and received medical assessment of the surgical success (documented absence of sperm), plus condom in male subject
  * Female partner is surgically sterilised (including hysterectomy), plus condom in male subject
  * Female partner is postmenopausal, defined as no menses for at least 1 year without an alternative medical cause, plus condom in male subject Alternatively, true abstinence is acceptable, if it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active, but becomes active with their partner, they must comply with the contraceptive requirements detailed above.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)(subjects with heart rate values between 45 and 50 bpm may be enrolled in case they have a normal thyroid function, no clinical symptoms associated with the bradycardia and no apparent signs of other diseases causing bradycardia such as hypothyroidism)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Major surgery (major according to the investigator's assessment) performed within 3 months prior to screening or planned after screening during the study, e.g. hip replacement
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 183 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in serum over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 183 days
Maximum measured concentration of the analyte in serum (Cmax) | up to 183 days

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com